CLINICAL TRIAL: NCT01477437
Title: Development and Evaluation of an Internet-based Educational Program to Promote Self- Management for Teens With Hemophilia
Brief Title: Internet-based Educational Program to Promote Self-Management for Teens With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinical Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000023483
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Hemophilia A
Keywords: teens; adolescents; Internet intervention; Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (experimental) Group (Experimental)
  Interventions: Other: Teens Taking Charge: Managing Hemophilia Online- Online self-management intervention
- Control group (No Intervention)

INTERVENTIONS:
Other: Teens Taking Charge: Managing Hemophilia Online- Online self-management intervention — The content will be delivered on a password-protected website, as part of the "About Kids Health" interface developed and maintained at the Hospital for Sick Children, Toronto, Canada. The website has been developed as eight discrete educational modules for adolescents. Each module takes approximately 30 to 45 minutes to complete. Content has been written and reviewed by experts from comprehensive hemophilia care clinics across Canada (physicians, nurses, physiotherapists and social workers) and edited by a medical writer to ensure that it is written at the suggested grade 6 reading level for patient education materials. Content has been written in English and will be translated into French prior to program launch. The format is geared towards adolescents and includes narratives with video components and interactive illustrations. In addition, each module will have quiz questions with real-time feedback to promote interactivity and knowledge retention.
  Arms: Intervention (experimental) Group

SUMMARY:
In summary, there is a clear need to improve knowledge and self-management skills in adolescents with hemophilia. To date, there are no published accounts of self-management programs for this population. Evidence from other chronic diseases that affects teens suggests that by developing an interactive Internet-based program, the investigators can meet the educational needs of adolescents with hemophilia and improve their ability to manage their hemophilia. In the long-term, improved self-management should result in a smoother and more successful transition to adult care and improve patient outcomes.

DETAILED DESCRIPTION:
The overall aim of this program of research is to develop and evaluate the "Teens Taking Charge: Managing Hemophilia Online" Internet intervention that will help adolescents with hemophilia to better understand and manage their disease independently. This program is modeled after Dr. Stinson's similar successful internet self-management program developed for youth with arthritis.

This program is being developed and evaluated using a sequential, phased approach. The first phase of this project has determined the self-management and transitional care needs of adolescents with hemophilia. Currently, in Phase 2A, we are developing the website with the content based on the findings from the Phase 1 needs assessment. We propose the current study to conduct usability testing (Phase 2B) to make sure it is easy to use and understand, and is efficient and satisfying to complete. Subsequently, we will assess the feasibility of the program and the outcomes from the use of the site in a randomized controlled trial (RCT) pilot study (Phase 3). This will enable us to determine an appropriate sample size for the future mixed controlled trial. Phases 2B and 3 are the focus of this proposal. Phase 4 will be a multicentre randomized controlled trial to assess outcomes for teens that complete the intervention as compared to those of an attention control group. This randomized controlled trial controlled trial will include all interested pediatric hemophilia treatment centres across Canada.

We hypothesize that adolescents with hemophilia who complete the "Teens Taking Charge: Managing Hemophilia Online" Internet intervention will demonstrate: increased hemophilia specific knowledge, increased self-efficacy, improved health-related quality of life (HRQL) and decreased stress prior to transition to adult health care.

ELIGIBILITY:
Inclusion Criteria:

* age 13-18
* diagnosis of mild, moderate or severe hemophilia A or B
* be able to speak and read English or French.
* must have access to the Internet at home

Exclusion Criteria

* cognitive impairments
* haematologist feels that they have a significant medical or psychiatric condition that will impact their participation
* don't have access to the internet.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Disease-specific knowledge gained | Baseline
  assessed by pre and post-assessment of the "Hemophilia Knowledge Questionnaire". This novel tool will be developed by investigators based on core content deemed important by hemophilia care providers and be reviewed for face validity by the Hemophilia Care Teams in both study centers and by a National panel of reviewers prior to administration.
Disease-specific knowledge gained | Immediately post-intervention - 8 weeks
  assessed by pre and post-assessment of the "Hemophilia Knowledge Questionnaire". This novel tool will be developed by investigators based on core content deemed important by hemophilia care providers and be reviewed for face validity by the Hemophilia Care Teams in both study centers and by a National panel of reviewers prior to administration.

SECONDARY OUTCOMES:
Health-related Quality of Life (HRQL) | Baseline and immediately post-intervention - 8 weeks
  Assessed pre and post intervention using the CHOK-LAT (Canadian Hemophilia Outcomes- Kids' Life Assessment Tool). This 35 item tool was developed at the Hospital for Sick Children and has been shown to be reliable and valid in assessing HRQL in children and adolescents with hemophila
Self-efficacy (Generalised Self-Efficacy-Sherer Scale) | Baseline and immediately post-intervention - 8 weeks
  This tool measures self efficacy. The 17-item scale was originally developed by Sherer and modified by Bosscher and Smit to include 12 items in three sub-scales (initiative, effort and persistence). This scale has been validated and found to be reliable in diverse populations. Although not validated specifically in adolescents, it has been used to study this population.
Preparedness for Transition | Baseline and immediately post-intervention - 8 weeks
  Measured using questionnaire developed by the John Hopkins Adult Cystic Fibrosis Program in a survey analyzing patient attitudes towards transition. The questions from this questionnaire have already been used in transition studies focused adolescents with hemophilia
Impact of the program | Baseline and immediately post-intervention - 8 weeks
  Will be measured in the intervention group only using the HEI-Q (Health Information Impact Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Breakey VR, Ignas DM, Warias AV, White M, Blanchette VS, Stinson JN. A pilot randomized control trial to evaluate the feasibility of an Internet-based self-management and transitional care program for youth with haemophilia. Haemophilia. 2014 Nov;20(6):784-93. doi: 10.1111/hae.12488. Epub 2014 Oct 14. PMID 25311370